CLINICAL TRIAL: NCT04199884
Title: Online Psychoeducation for Intolerance of Uncertainty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: Mary Oglesby Shapiro (Unknown)
Responsible Party: Principal Investigator, Norman Schmidt, Distinguished Research Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Oglesby02
Record Dates: First submitted 2019-12-12; First posted 2019-12-16 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Intolerance of Uncertainty; Anxiety
Keywords: Intolerance of Uncertainty; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active IU-focused Psychoeducation Intervention (Experimental)
  Interventions: Behavioral: Active IU-focused Psychoeducation Intervention
- Health-focused Psychoeducation Intervention (Active Comparator)
  Interventions: Behavioral: Health-focused Psychoeducation Intervention

INTERVENTIONS:
Behavioral: Active IU-focused Psychoeducation Intervention — This paradigm was an IU-focused psychoeducation intervention wherein participants were provided psychoeducation about the nature of IU and anxiety, given strategies to cope with fear of uncertainty, and provided examples and information as to how they can expose themselves to uncertainty.
  Arms: Active IU-focused Psychoeducation Intervention
Behavioral: Health-focused Psychoeducation Intervention — This intervention is a health-focused psychoeducation intervention wherein participants learn ways to engage in healthy behaviors, such as getting adequate sleep, eating healthier, and exercising regularly.
  Arms: Health-focused Psychoeducation Intervention

SUMMARY:
Randomized control trial examining the efficacy of an online intolerance of uncertainty focused psychoeducation intervention.

DETAILED DESCRIPTION:
Randomized control trial examining the efficacy of an online intolerance of uncertainty (IU) focused psychoeducation intervention among females elevated in IU.

ELIGIBILITY:
Inclusion Criteria:

* Elevated intolerance of uncertainty at baseline

Exclusion Criteria:

* Patients would be excluded if they endorsed suicidal ideation/intent that required hospitalization.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Intolerance of Uncertainty (IIU) | Baseline to one-month follow-up
  Change IU across time
Beck Anxiety Inventory | Baseline to one-month follow-up
  Change in beck anxiety inventory scores across time

CONTACTS AND LOCATIONS:
Locations (1):
- Anxiety and Behavioral Health Clinic, Tallahassee, Florida, United States